CLINICAL TRIAL: NCT07042295
Title: A Randomized Phase II Study of Amivantamab (JNJ-61186372) and Hyaluronidase (rHuPH20) Versus Cetuximab in Immunocompromised Participants With Recurrent Inoperable or Metastatic Cutaneous Squamous Cell Carcinoma
Brief Title: Treatment With Amivantamab and Hyaluronidase or Cetuximab for Advanced Skin Cancer in People With a Weakened Immune System
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-04318; NCI-2025-04318 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SN2426 (Other: SWOG); SN2426 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2025-06-27; First posted 2025-06-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Locally Recurrent Skin Squamous Cell Carcinoma; Metastatic Skin Squamous Cell Carcinoma
MeSH Terms: interventions — amivantamab; Hyaluronoglucosaminidase; Specimen Handling; Cetuximab; (225)Ac-DOTA-c(RGDyK); Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (amivantamab and hyaluronidase) (Experimental): Patients receive amivantamab and hyaluronidase SC over at least 5 minutes on days 1, 8, 15 and 22 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection on study and CT scan and/or MRI throughout the study.
  Interventions: Drug: Amivantamab and Recombinant Human Hyaluronidase; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm II (cetuximab) (Active Comparator): Patients receive cetuximab IV over 60-120 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection on study and CT and/or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Cetuximab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Amivantamab and Recombinant Human Hyaluronidase — Given SC
  Other Names: Amivantamab + Recombinant Human Hyaluronidase; Amivantamab and Hyaluronidase; Amivantamab Plus Recombinant Human Hyaluronidase; Amivantamab with Recombinant Human Hyaluronidase; Amivantamab-Recombinant Human Hyaluronidase; Amivantamab/Recombinant Human Hyaluronidase
  Arms: Arm I (amivantamab and hyaluronidase)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm II (cetuximab)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial compares the effect of amivantamab and hyaluronidase to cetuximab for the treatment of skin (cutaneous) squamous cell carcinoma that has come back after a period of improvement and has not spread to other parts of the body (locally recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Amivantamab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Hyaluronidase is an endoglycosidase. It helps to keep amivantamab in the body longer, so that the medications will have a greater effect. Cetuximab is in a class of medications called monoclonal antibodies. It binds to a protein called EGFR, which is found on some types of cancer cells. This may help keep cancer cells from growing. Giving amivantamab and hyaluronidase may be as effective as cetuximab for the treatment of locally recurrent or metastatic cutaneous squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and preliminary efficacy of amivantamab monotherapy in patients with locoregionally incurable or metastatic cutaneous squamous cell carcinoma and an active immunosuppressed condition. (Cohort A) II. To compare progression-free survival (PFS) of amivantamab monotherapy versus cetuximab monotherapy in patients with locoregionally incurable or metastatic cutaneous squamous cell carcinoma and an active immunosuppressed condition. (Cohort B)

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities in each cohort and treatment arm.

II. To estimate confirmed objective response rate (ORR) (ORR, confirmed complete and partial responses by Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1) in each cohort and treatment arm.

III. To estimate duration of objective response, time to progression, time to next treatment, and overall survival in each cohort and treatment arm.

IV. To estimate ORR and progression free survival (PFS) in each cohort and treatment arm in subgroups defined by reason for immunosuppression: transplant, autoimmune disease, hematologic malignancy, or other reason.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients in cohort A are assigned to arm I, patients in cohort B are randomized to arm I or II.

ARM I: Patients receive amivantamab and hyaluronidase subcutaneously (SC) over at least 5 minutes on days 1, 8, 15 and 22 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection on study and computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the study.

ARM II: Patients receive cetuximab intravenously (IV) over 60-120 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection on study and CT and/or MRI throughout the study.

After completion of study treatment, patients are followed up, per the treating investigator, for up 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically proven diagnosis of cutaneous squamous cell carcinoma based on pathology from original diagnosis or from a metastatic/recurrent lesion
* Participants must have measurable or non-measurable disease per RECIST 1.1 and must have their disease assessed by CT of chest/abdomen/pelvis (with contrast unless contraindicated) within 28 days prior to registration for measurable disease or within 42 days prior to registration for non-measurable disease. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form (RECIST 1.1). Any lesions assessed using a non-diagnostic positron emission tomography (PET)/CT of chest/abdomen/pelvis will be considered non-measurable lesions. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration to be considered measurable

  * NOTE: All diseases must be assessed and documented on the baseline tumor assessment form
* Participants with exclusively locally recurrent disease must have either a contraindication to surgical treatment of lesions (i.e., complete resection is not possible or not expected to be clinically beneficial or resection conferring significant cosmetic or functional concerns) or have refused surgical or radiation treatment
* Participants must be immunocompromised, defined as below. For cases where there is a lack of clarity, it is highly recommended study teams reach out to Drs. Swiecicki and Geiger for discussion:

  * An active diagnosis of either chronic lymphocytic leukemia (CLL) or acute leukemia, regardless of whether actively receiving therapy OR
  * A diagnosis of lymphoma or multiple myeloma either on antineoplastic therapy, or within 6 months after therapy completion OR
  * Recipient of an organ transplant (excluding corneal transplants or lung transplants)

    * If a transplant patient, documentation from the patient's transplant physician confirming that the patient's allograft is stable. Documentation must be dated within 180 days of registration OR
  * Autoimmune disease under active treatment with an immunosuppressive medication (as defined below)

    * Autoimmune diseases include but are not limited to: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, myasthenia gravis, Guillain-Barre syndrome, autoimmune hepatitis, scleroderma, primary biliary cirrhosis, pemphigus, and bullous pemphigoid

      * Vitiligo, psoriasis, type 1 diabetes mellitus, hypothyroidism, or resolved childhood asthma/atopy are not eligible diagnoses
    * Immunosuppressant medications include the following:

      * Tumor necrosis factor (TNF) inhibitors (adalimumab, certolizumab, etanercept, golimumab, and infliximab)
      * Interleukin inhibitors (anakinra, ustekinumab, secukinumab, sarilumab, siltuximab, sulfasalazine, tildrakizumab, tocilizumab, chloroquine, and hydroxychloroquine)
      * Janus kinase (JAK) inhibitors (baricitinib, filgotinib, and tofacitinib)
      * Calcineurin inhibitors (cyclosporine and tacrolimus)
      * Metabolic inhibitors (azathioprine, leflunomide, mercaptopurine, methotrexate)
      * mTOR (mammalian target of rapamycin) inhibitors (sirolimus [rapamycin], everolimus, and zotarolimus)
      * Inosine monophosphate dehydrogenase inhibitors (mycophenolate)
      * Phosphodiesterase inhibitors (apremilast)
      * B cell inhibitors (rituximab)
      * T cell inhibitors (abatacept)
      * Glucocorticoids
    * Active treatment is defined as current use of any one or more of the following:

      * Oral glucocorticoid therapy (Prednisone equivalent > 10 mg/day) for 30 days prior to registration
      * Oral or subcutaneous immunosuppressive therapy for 90 days or more prior to registration
      * Two or more doses of intravenous non corticosteroid immunosuppressant within 90 days prior to registration
* Participants with treated brain metastases must show no evidence of progression on follow-up brain imaging after central nervous system (CNS)-directed therapy
* Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease must not require immediate CNS specific treatment at the time of study registration or anticipated during the first cycle of therapy
* Participants must not have had prior treatment with cetuximab or another EGFR inhibitor within the last 365 days
* Participant must be ≥ 18 years old at the time of registration
* Participant must have Zubrod Performance Status of 0-2
* Participant must have a complete medical history and physical exam within 28 days prior to registration
* Leukocytes ≥ 3 x 10^3/uL (within 14 days prior to registration)
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 14 days prior to registration)
* Platelets ≥ 100 x 10^3/uL (within 14 days prior to registration)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN (within 14 days prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 × institutional ULN with the exception of subjects with documented liver metastases: AST and/or ALT ≤ 5.0 x institutional ULN (within 14 days prior to registration)
* Participants must have a measured OR calculated creatinine clearance ≥ 30 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 14 days prior to registration
* Participants must not have an active or past medical history of interstitial lung disease (ILD)/pneumonitis, including drug-induced or radiation ILD/pneumonitis
* Participants must not have a history of lung transplantation
* Participants must not have a history of pulmonary graft versus host disease (GVHD)
* Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* Participants with a history human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* Participants with a history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants must not have an uncontrolled illness, including but not limited to:

  * Ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting study treatment])
  * Active bleeding diathesis
  * Any ophthalmologic condition that is clinically unstable
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped) due to known toxicities of amivantamab. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen. Participants must agree not to donate ova or sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study treatment. For female participants of childbearing potential, a negative pregnancy test is required within 72 hours prior to registration
* Participants must be offered the opportunity to participate in specimen banking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-10-25 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity of interest (cohort A) | Up to completion of the first cycle (cycle length = 28 days)
  Defined as grade 3 or 4 skin rash that does not recover within 14 days, grade 3 or 4 non-hematologic toxicity that does not recover within 7 days, grade 4 hematologic toxicity including febrile neutropenia or organ transplant failure (for transplant patients only).
Progression free survival (PFS) (cohort B) | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, up to 3 years

SECONDARY OUTCOMES:
Organ rejection | Up to 5 years
  Will be monitored for participants with prior organ transplants.
Overall survival (OS) | From date of registration to date of death due to any cause, up to 5 years
  Will estimate OS by cohort and treatment arm and within subgroups using the method of Kaplan-Meier. OS will be compared between arms using an un-stratified log-rank test. The hazard ratio and 95% confidence interval from an un-stratified Cox regression model with treatment as the only covariate will be descriptively reported for OS.
PFS | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, up to 5 years
  Will estimate PFS by cohort and treatment arm and within subgroups using the method of Kaplan-Meier.
Time to next treatment | Up to 3 years
  will be estimated using cumulative incidence curves with death before event accounted for as a competing event.
Time to progression | Up to 3 years
  will be estimated using cumulative incidence curves with death before event accounted for as a competing event.
Duration of objective response | Up to 5 years
  Will be estimated using cumulative incidence curves with death before event accounted for as a competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Swiecicki, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- SWOG, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm